CLINICAL TRIAL: NCT00803972
Title: A Phase I, Randomized, Dose-Ranging, Pharmacokinetic, Glucodynamic, Safety, and Tolerability Study of SC Administered Humulin R and Humalog With or Without Recombinant Human Hyaluronidase (rHuPH20) in Healthy Volunteers
Brief Title: Dose-Ranging, Pharmacokinetic (PK), Glucodynamic (GD), Safety and Tolerability Study of Subcutaneously (SC) Administered Humulin R and Humalog With or Without rHuPH20
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HZ2-08-04
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: Humalog; Humulin R; rHuPH20; Hylenex
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Stage 1: 3 U insulin plus rHuPH20 (Experimental): Participants will receive 3 Units (U) of regular insulin (100 U/milliliter [mL]), coadministered with sequential concentrations of 0, 1.25, 5, 10, 20, and 80 micrograms (μg)/mL recombinant human hyaluronidase (rHuPH20).
  Interventions: Drug: rHuPH20; Drug: Insulin Human Injection
- Stage 1: 12 U insulin plus rHuPH20 (Experimental): Participants will receive 12 U of regular insulin (100 U/mL), coadministered with sequential concentrations of 0, 1.25, 5, 10, 20, and 80 μg/mL rHuPH20.
  Interventions: Drug: rHuPH20; Drug: Insulin Human Injection
- Stage 2: insulin plus rHuPH20 (Experimental): Participants will receive 6, 12, and 24 U regular insulin (100 U/mL) in a randomly assigned order, with each insulin dose administered once with and once without 5 μg/mL rHuPH20.
  Interventions: Drug: rHuPH20; Drug: Insulin Human Injection
- Stage 3: 1.5 U insulin lispro plus rHuPH20 (Experimental): Participants will receive 1.5 U of insulin lispro (50 U/mL), coadministered with sequential concentrations of 0, 0.0625, 0.3125, 1.25, 5, and 20 μg/mL rHuPH20.
  Interventions: Drug: rHuPH20; Drug: Insulin Lispro Injection
- Stage 3: 6 U insulin lispro plus rHuPH20 (Experimental): Participants will receive 6 U of insulin lispro (50 U/mL), coadministered with sequential concentrations of 0, 0.0625, 0.3125, 1.25, 5, and 20 μg/mL rHuPH20.
  Interventions: Drug: rHuPH20; Drug: Insulin Lispro Injection
- Stage 4: 95 U/mL insulin lispro plus 5 μg/mL rHuPH20 (Experimental): Participants will receive 95 U/mL insulin lispro, administered once with and once without 5 μg/mL rHuPH20. At each insulin lispro concentration, participants will receive 2, 6, and 20 U lispro.
  Interventions: Drug: rHuPH20; Drug: Insulin Lispro Injection
- Stage 4: 50 U/mL insulin lispro plus 5 μg/mL rHuPH20 (Experimental): Participants will receive 50 U/mL insulin lispro, administered once with and once without 5 μg/mL rHuPH20. At each insulin lispro concentration, participants will receive 2, 6, and 20 U lispro.
  Interventions: Drug: rHuPH20; Drug: Insulin Lispro Injection
- Stage 4: 25 U/mL insulin lispro plus 5 μg/mL rHuPH20 (Experimental): Participants will receive 25 U/mL insulin lispro, administered once with and once without 5 μg/mL rHuPH20. At each insulin lispro concentration, participants will receive 2, 6, and 20 U lispro.
  Interventions: Drug: rHuPH20; Drug: Insulin Lispro Injection

INTERVENTIONS:
Drug: rHuPH20 — recombinant human hyaluronidase PH20
Drug: Insulin Human Injection — injection
  Other Names: Humulin® R
  Arms: Stage 1: 12 U insulin plus rHuPH20; Stage 1: 3 U insulin plus rHuPH20; Stage 2: insulin plus rHuPH20
Drug: Insulin Lispro Injection — injection
  Other Names: Humalog®
  Arms: Stage 3: 1.5 U insulin lispro plus rHuPH20; Stage 3: 6 U insulin lispro plus rHuPH20; Stage 4: 25 U/mL insulin lispro plus 5 μg/mL rHuPH20; Stage 4: 50 U/mL insulin lispro plus 5 μg/mL rHuPH20; Stage 4: 95 U/mL insulin lispro plus 5 μg/mL rHuPH20

SUMMARY:
This is a single center, Phase I, open-label, single-blind (subjects blinded to the contents of each injection), 4 stage study designed to determine the PK, GD, safety, tolerability, and optimal ratio of rHuPH20 administered with fixed Humulin R or Humalog doses in healthy subjects.

DETAILED DESCRIPTION:
Subjects will be enrolled in one of four sequential study stages. In each stage, a euglycemic clamp procedure will be used to control plasma glucose levels. Blood samples will be collected over an 8-hour time period after insulin administration (either Humulin R or Humalog) to analyze insulin and glucose levels using fully validated methods. Glucose infusion rates (GIR) will be recorded throughout the study period. The study is single-blind, with study subjects blinded as to the contents of each injection.

Determine the pharmacokinetics (PK) and optimum ratio of rHuPH20:insulin when a range of rHuPH20 dose ratios are administered subcutaneously (SC) with fixed doses of Humulin R, by determining Tmax, Cmax, AUCs, and relative bioavailability based on serum insulin concentrations collected at specified time points (Stage 1).

Determine if different concentrations of Humulin R impact the PK and minimal rHuPH20 dose necessary to achieve full insulin PK effect over a representative range of typical prandial SC Humulin R doses using the rHuPH20:insulin ratio identified in Stage 1 (Stage 2).

Determine the PK and optimum ratio of rHuPH20:insulin when a range of rHuPH20 dose ratios are administered SC with fixed doses of Humalog, by determining Tmax, Cmax, AUCs, and relative bioavailability based on serum insulin concentrations collected at specified time points (Stage 3).

Determine if different concentrations of Humalog impact the PK and minimal rHuPH20 dose necessary to achieve full insulin PK effect over a representative range of typical prandial SC Humalog doses using the rHuPH20:insulin ratio identified in Stage 3 (Stage 4).

Evaluate the safety and local tolerability of the SC injection at various rHuPH20, Humulin R, and Humalog doses (Stages 1 - 4).

Assess the glucodynamics (GD) of the SC injection of various rHuPH20, Humulin R, and Humalog doses (Stages 1 - 4).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination (PE), including blood pressure (BP) and heart rate (HR), 12-lead electrocardiogram (ECG) and clinical laboratory tests specified in these eligibility criteria).
* BMI between 18-28 kg/m2, inclusive.
* Total body weight >70 kg (154 lb) for men and 46 kg (101 lb) for women.
* Subject willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including adequate venous access.
* Vital signs (BP, HR, temperature, respiratory rate) within normal range or, if out of range, assessed by the Principal Investigator (PI) as not clinically significant (NCS) and mutually agreed by both PI and the Sponsor's medical monitor that the subject need not be excluded from the study for this abnormal value.
* Within 14 days before the first injection: metabolic panel (e.g., sodium, potassium, chloride, bicarbonate, BUN (blood urea nitrogen), creatinine, glucose, calcium, AST (aspartate transaminase [SGOT]), ALT (alanine transaminase [SGPT]), alkaline phosphatase, total bilirubin, albumin, cholesterol, lipids, amylase and total protein) and complete blood count (CBC) within the laboratory normal reference range or, if out of range, assessed by the PI as NCS and mutually agreed by both PI and the Sponsor's medical monitor that the subject need not be excluded from the study for this laboratory value.
* Fasting plasma glucose level within the range of 60 to 100 mg/dL, inclusive, within 30 minutes of the first euglycemic clamp.
* A negative serum pregnancy test (if female of childbearing potential) within 14 days of study drug injection.
* Female subjects of childbearing potential must agree to be practicing effective birth control or abstinence currently and agree to continue to do so for the duration of their time on study.
* Decision-making capacity and willingness and ability to comply with the requirements for full completion of the study.
* Signed, written IRB-approved informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, oncologic, or neurologic (to include history of seizures) disease; hypoglycemic episodes; intercurrent illness (such as influenza); or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). Clinical significance to be determined by the PI.
* Known history of diabetes mellitus or gestational diabetes.
* Known allergy to hyaluronidase or any other ingredient in the study drug.
* Positive HIV 1 and HIV 2 (human immunodeficiency virus) antibody test, hepatitis B (anti-HBsAg) or hepatitis C (anti-HCV) antibody test.
* Any history or evidence of alcohol or drug abuse.
* History or evidence of use of any tobacco- or nicotine-containing product within 6 months of screening, screening quantitative urine nicotine concentration >50 ng/mL, or screening serum cotinine concentration of > 20 ng/mL.
* Use of drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action or glucose utilization.
* Donation of blood in excess of 500 mL within 56 days before dosing.
* Failure to limit alcohol consumption and refrain from exercise within 48 hours before each injection.
* Participation in a study of any investigational drug or device 30 days before enrollment in this study.
* The subject is unfit for the study in the opinion of the investigator.
* Women who are pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08-28 (Actual); Study Completion 2009-08-28 (Actual)

PRIMARY OUTCOMES:
Insulin AUC | 0 to 60 minutes

SECONDARY OUTCOMES:
Other insulin PK, GD and safety outcomes | Day of each injection and 7 days after final dose

CONTACTS AND LOCATIONS:
Overall Officials: Jolene K Berg, MD, Principal Investigator — dgd Research, Inc.
Locations (1):
- dgd Research, Inc., San Antonio, Texas, United States